CLINICAL TRIAL: NCT02425202
Title: Ketamine Infusion for Pediatric Patients With Obstructive Sleep Apnea Syndrome After Tonsillectomy: A Randomized Controlled Trial
Brief Title: Ketamine Infusion for Pediatric Patients With Obstructive Sleep Apnea Syndrome (OSAS) After Tonsillectomy
Acronym: KOSATA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2013:163
Record Dates: First submitted 2015-04-14; First posted 2015-04-23 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-05

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: pediatric; obstructive sleep apnea; tonsillectomy; analgesia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Agnosia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine infusion (Active Comparator): Ketamine infusion at 0.1 mg/kg/hr up to maximum of 10 mg/hr
  Interventions: Drug: Ketamine
- Saline infusion (Placebo Comparator): Saline infusion
  Interventions: Other: Saline infusion

INTERVENTIONS:
Drug: Ketamine — Post-operative continuous infusion until 0600 the next day
  Other Names: Ketalar
  Arms: Ketamine infusion
Other: Saline infusion — Post-operative continuous infusion until 0600 the next day
  Other Names: Placebo comparator
  Arms: Saline infusion

SUMMARY:
The study will evaluate the post-operative morphine-sparing effect, pain reduction, and side effects of a continuous ketamine infusion after tonsillectomy in pediatric patients.

DETAILED DESCRIPTION:
Eligible pediatric patients that are undergoing tonsillectomy for sleep-disordered breathing or obstructive sleep apnea AND are to be admitted into a monitored setting will be recruited for this study. They will be randomized into two groups:1) Control group receiving continuous infusion of saline (placebo) and 2) Study group receiving continuous infusion of low-dose ketamine at 0.1 mg/kg/hr. Both patients will receive scheduled oral acetaminophen and rescue intravenous morphine as required. The infusions will be stopped at 0600 the next morning. Morphine requirements, pain scores at selected times, central nervous system side effects, and adverse cardiorespiratory events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring tonsillectomy for diagnosis of sleep disordered breathing/obstructive sleep apnea that will be admitted for overnight cardiorespiratory monitoring, based on positive polysomnography test, positive nocturnal home oximetry, or strong signs/symptoms of OSAS

Exclusion Criteria:

* Patients with significant developmental delay, abnormal airway anatomy, significant co-morbidities such as cardiac disorders, respiratory disorders, neurological disorders, anad renal disorders.
* Previous reaction to study medications.
* Postoperative bleeding within the first 24 hours
* Refusal to be involved in the study..

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2014-12; Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Measurement of post-operative opioid requirements after tonsillectomy in obstructive sleep apnea (OSA) patients | 24 hrs
  Influence of low-dose continuous ketamine infusion on post-operative opioid requirements after tonsillectomy in OSA patients.

SECONDARY OUTCOMES:
Documentation of respiratory morbidity after tonsillectomy in OSA patients | 24 hrs
  Influence of low-dose ketamine infusion on respiratory morbidity after tonsillectomy in OSA patients

CONTACTS AND LOCATIONS:
Overall Officials: Harley Wong, MD, FRCPC, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Center, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brown KA. Outcome, risk, and error and the child with obstructive sleep apnea. Paediatr Anaesth. 2011 Jul;21(7):771-80. doi: 10.1111/j.1460-9592.2011.03597.x. Epub 2011 May 3. PMID 21539679
- [Result] Alexander NS, Schroeder JW Jr. Pediatric obstructive sleep apnea syndrome. Pediatr Clin North Am. 2013 Aug;60(4):827-40. doi: 10.1016/j.pcl.2013.04.009. PMID 23905822
- [Result] Bhattacharjee R, Kheirandish-Gozal L, Spruyt K, Mitchell RB, Promchiarak J, Simakajornboon N, Kaditis AG, Splaingard D, Splaingard M, Brooks LJ, Marcus CL, Sin S, Arens R, Verhulst SL, Gozal D. Adenotonsillectomy outcomes in treatment of obstructive sleep apnea in children: a multicenter retrospective study. Am J Respir Crit Care Med. 2010 Sep 1;182(5):676-83. doi: 10.1164/rccm.200912-1930OC. Epub 2010 May 6. PMID 20448096
- [Result] Petrenko AB, Yamakura T, Baba H, Shimoji K. The role of N-methyl-D-aspartate (NMDA) receptors in pain: a review. Anesth Analg. 2003 Oct;97(4):1108-1116. doi: 10.1213/01.ANE.0000081061.12235.55. PMID 14500166
- [Result] Baugh RF, Archer SM, Mitchell RB, Rosenfeld RM, Amin R, Burns JJ, Darrow DH, Giordano T, Litman RS, Li KK, Mannix ME, Schwartz RH, Setzen G, Wald ER, Wall E, Sandberg G, Patel MM; American Academy of Otolaryngology-Head and Neck Surgery Foundation. Clinical practice guideline: tonsillectomy in children. Otolaryngol Head Neck Surg. 2011 Jan;144(1 Suppl):S1-30. doi: 10.1177/0194599810389949. PMID 21493257